CLINICAL TRIAL: NCT05288907
Title: SOOTHER Trial: Study of an Over-the-Counter Ointment to Treat Rectal Itch
Brief Title: SOOTHER Trial to Treat Rectal Itch
Status: Completed | Type: Observational
Sponsor: Bell International Laboratories (Industry)
Responsible Party: Sponsor
Other Study IDs: 20181914
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Pruritus Ani
Keywords: Pruritus ani; rectal itch; anal itch
MeSH Terms: conditions — Pruritus Ani

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pruritus ani patients: Adult patients with pruritus ani (rectal itch) treated with lidocaine ointment
  Interventions: Drug: Lidocaine Ointment

INTERVENTIONS:
Drug: Lidocaine Ointment — Composite over-the-counter lidocaine ointment administered twice daily for 2 weeks.

SUMMARY:
Longitudinal, observational, single-arm trial of a novel, composite Lidocaine ointment to treat rectal itch (pruritus ani)

ELIGIBILITY:
Inclusion Criteria:

* Presence of pruritus ani (anal itch/discomfort) for at least 2 weeks, and a compatible physical exam.

Exclusion Criteria:

* Inability to understand informed consent, history of inflammatory bowel disease, known venereal disease, or immunodeficiency disease, history of or current anal or perianal abscess, anal or rectal surgery within the past 12 weeks, pregnancy or breastfeeding female, or signs of other rectal diseases such as anorectal fistula, infection, perianal eczema or tumors.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with pruritus ani (anal itch/discomfort)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-08-13 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Symptom assessment | 2 weeks
  SOOTHER Symptom assessment at 2 weeks rated on a 5-point analog scale, with 5 being the worst
Visual ano-rectal exam | 2 weeks
  Visual ano-rectal exam assessment at 2 weeks rated on a 5-point analog scale, with 5 being the worst.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Saremi, Principal Investigator — Bell International Laboratories
Locations (1):
- Minnesota Gastroenterology, Plymouth, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Felemovicius I, Ganz RA, Saremi M, Christopfel W. SOOTHER TRIAL: Observational study of an over-the-counter ointment to heal anal itch. Front Med (Lausanne). 2022 Sep 14;9:890883. doi: 10.3389/fmed.2022.890883. eCollection 2022. PMID 36186810